CLINICAL TRIAL: NCT01064453
Title: Angeliq Regulatory Post Marketing Surveillance
Acronym: Angeliq rPMS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14841; AQ0710KR (Other: company internal)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Postmenopausal Period; Osteoporosis, Postmenopausal
Keywords: Menopause; Menopausal symptoms; Prevention of osteoporosis in menopausal women; Estrogen deficiency symptoms; Hormone replacement therapy
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — estradiol-drospirenone combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: E2/DRSP (Angeliq, BAY86-4891)

INTERVENTIONS:
Drug: E2/DRSP (Angeliq, BAY86-4891) — Take one tablet daily, continuously

SUMMARY:
Angeliq regulatory Post-Marketing Surveillance (PMS) is to get data about safety and efficacy in real practice for the indication approved by Korea Food and Drug Administration (KFDA). This is non-interventional , prospective, multi-center study.Target number of patients is 4500.

ELIGIBILITY:
Inclusion Criteria:

* Hormone replacement therapy for estrogen deficiency symptoms in postmenopausal women more than 1 year postmenopause
* Prevention of osteoporosis in postmenopausal women at high risk of future fractures who are intolerant of, or contraindicated for, other medicinal products approved for the prevention of osteoporosis

Exclusion Criteria:

* Undiagnosed genital bleeding
* Known, past or suspected cancer of the breast
* Known or suspected estrogen-dependent malignant tumors (e.g. endometrial cancer)
* Untreated endometrial hyperplasia
* Previous idiopathic or current venous thromboembolism (e.g. deep venous thrombosis, pulmonary embolism)
* Active or recent arterial thromboembolic disease (e.g. angina, myocardial infarction)
* Acute liver disease, or a history of liver disease as long as liver function tests have failed to return to normal
* Porphyria
* Severe renal insufficiency or acute renal failure
* Known hypersensitivity to the active substances or to any of the excipients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean women who take Angeliq for postmenopausal symptoms or/and prevention of osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 4078 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Adverse event collection | At each visit of patient during observational period (6 months)

SECONDARY OUTCOMES:
Improvement of menopausal symptoms | After 6 months or at discontinuation of Angeliq (At earlier point)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea